CLINICAL TRIAL: NCT05883878
Title: Innovative Approaches for Personalised Cardiovascular Prevention: Multicenter Randomised Controlled Study and Multidisciplinary Evaluation for a National Health Service (NHS) Implementation
Brief Title: Innovative Approaches for Personalised Cardiovascular Prevention
Acronym: INNOPREV
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Collaborators: University Of Perugia (Other); Policlinic Hospital "G. Rodolico" (Other); Azienda Ospedaliera Universitaria Policlinico Paolo Giaccone Palermo (Other)
Responsible Party: Principal Investigator, Boccia Stefania, Full Professor of Hygiene and Preventive Medicine, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 5506
Record Dates: First submitted 2023-05-17; First posted 2023-06-01 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Cardiovascular Diseases
Keywords: Coronary Artery Disease (CAD)
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Artery Disease | interventions — Wearable Electronic Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Standard of Care (No Intervention): Participants will receive traditional lifestyle advices in order to reduce the risk.
- Genetic testing - PRS (Experimental): Participants will receive the information of the genetic cardiovascular risk (PRS) and personalized advices.
  Interventions: Genetic: PRS
- Digital intervention - app and wearable device (Experimental): Participants will receive an app and a wearable device for the evaluation of various parameters.
  Interventions: Device: Digital app and wearable device
- Digital intervention and genetic testing - PRS (Experimental): Participants will receive both app and wearable device and PRS information
  Interventions: Genetic: PRS; Device: Digital app and wearable device

INTERVENTIONS:
Genetic: PRS — genetic test for the evaluation of PRS cardiovascular risk
  Arms: Digital intervention and genetic testing - PRS; Genetic testing - PRS
Device: Digital app and wearable device — a wearable device connected with its app
  Arms: Digital intervention - app and wearable device; Digital intervention and genetic testing - PRS

SUMMARY:
The goal of this clinical trial is to study innovative approaches for personalized primary preventive interventions for cardiovascular diseases (CVD) in the population. The main questions it aims to answer are:

* efficacy and safety of the intervention
* how to implement the interventions in the NHS

Participants will be randomized in one of the four parallel arms:

* standard of care;
* genetic testing for cardiovascular genetic risk (through the cardiovascular Polygenic Risk Score or PRS);
* digital intervention with a wearable device and its app;
* digital intervention and genetic testing (PRS)

The primary outcome we are going to evaluate is the efficacy of returning PRS information of CVD measured at baseline, alone or in combination with the use of a wearable device, on two endpoints: i) change in lifestyle pattern; ii) CVD risk profile modification. The postulated hypothesis is that the achievement of these endpoints is more likely in presence of at least one of the aforementioned interventions than among subjects who receive only traditional risk assessment at baseline, nor respect to subjects receiving traditional risk assessment plus adopting wearable devices.

DETAILED DESCRIPTION:
The trial will consist of four phases: an enrollment phase (T0), a disclosure visit three weeks later (T1), a follow-up visit five months after the disclosure visit (T2), and a final follow-up twelve months from enrollment (T3).

Once enrolled (T0), all participants will sign the informed consent form and undergo a comprehensive assessment, which includes:

* Completing a questionnaire on socioeconomic status, area of residence, and lifestyle, using the Life's Essential 8 tool [1]. The questionnaire will cover smoking status, alcohol consumption, dietary pattern, sleep pattern, and physical activity. Participants will be classified into favorable, intermediate, or unfavorable individual lifestyle patterns according to the Life's Essential 8 score.
* Blood analysis will be performed to evaluate the lipid profile, including total cholesterol, LDL cholesterol, HDL cholesterol, and triglycerides.

At T1, a disclosure visit will be conducted to explain the assigned lifestyle category, share the results of the blood tests, and provide information on the expected interventions based on the assigned group.

The questionnaire will be administered at T0, T2, and T3. Blood analysis and cardiovascular profile evaluation will be conducted at both T0 and T3

ELIGIBILITY:
Inclusion Criteria:

* high cardiovascular risk based on the SCORE 2 (between 2.5% and 10%)
* age between 40 and 69 years

Exclusion Criteria:

* diabetes.
* familiar hypercholesterolemia.
* established CVD.

Ages: 40 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1020 (Estimated)
Dates: Start 2023-07-24 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Change in the Lifestyle Category | 12 months
  The lifestyle category will be measured using the Life's Essential 8 tool. A change will be considered achieved if there is a shift towards a more favorable lifestyle category.
Modification of the Lipid Profile | 12 months
  We will evaluate whether there is a change in the lipid profile compared to the baseline value. The modification of the lipid profile can also be considered as an indicator of the modification of the cardiovascular risk profile measured with the SCORE 2 charts.

CONTACTS AND LOCATIONS:
Locations (1):
- Dipartimento Universitario di Scienze della Vita e Sanità Pubblica, Roma, Italia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lloyd-Jones DM, Allen NB, Anderson CAM, Black T, Brewer LC, Foraker RE, Grandner MA, Lavretsky H, Perak AM, Sharma G, Rosamond W; American Heart Association. Life's Essential 8: Updating and Enhancing the American Heart Association's Construct of Cardiovascular Health: A Presidential Advisory From the American Heart Association. Circulation. 2022 Aug 2;146(5):e18-e43. doi: 10.1161/CIR.0000000000001078. Epub 2022 Jun 29. PMID 35766027